CLINICAL TRIAL: NCT00054795
Title: Randomized Phase III Trial of Xcytrin® (Motexafin Gadolinium) Injection for the Treatment of Brain Metastases in Patients With Non-Small Cell Lung Cancer Undergoing Whole Brain Radiation Therapy
Brief Title: Study of Neurologic Progression With Motexafin Gadolinium and Radiation Therapy (SMART)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0211; NCT00066820 (obsolete NCT alias)
Record Dates: First submitted 2003-02-10; First posted 2003-02-13 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Metastases, Neoplasm
Keywords: Brain Neoplasms/radiotherapy; Neoplasms/complications/prevention & control,; Neuropsychological Tests,; Metalloporphyrins/therapeutic use,; Combined Modality Therapy,; Drug therapy,; Quality of Life,; Cranial Irradiation,; Radiotherapy/Targeted,; Prospective Studies,; Neoplasm Recurrence/Local,; Treatment Outcome; Brain metastases; Brain Neoplasms/secondary; Non-small cell lung cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Neoplasms; Neoplasm Recurrence, Local | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium

SUMMARY:
The primary purpose of the study is to determine if patients with brain metastases from non-small cell lung cancer treated with Motexafin Gadolinium and whole brain radiation therapy retain their neurologic function and ability to think for a longer time compared to patients treated with whole brain radiation therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with radiologically proven parenchymal brain metastases from histologically confirmed non-small cell lung cancer;
* KPS score of ≥70;
* Each patient must sign a study-specific Informed Consent form

Exclusion Criteria:

* Liver metastases;
* Extracranial metastases in two or more organs;
* Known leptomeningeal metastases or subarachnoid spread of tumor;
* Prior whole brain radiation;
* Plan to use radiosurgery or radiation boost after completion of WBRT;
* Planned chemotherapy during study treatment (prior and subsequent chemotherapy is allowed);
* Prior total resection of a single brain metastasis;
* Laboratory values as follows:

LDH > 1.3 x upper limit of normal (ULN); ANC < 1500 /mm³; Platelets < 50,000 /mm³; Creatinine > 2.0 mg/dL; AST or ALT > 2 x ULN; Total bilirubin > 2 x ULN;

* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550

CONTACTS AND LOCATIONS:
Locations (92):
- United States (44):
  - Phoenix, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Berkeley, California
  - Concord, California
  - Greenbrae, California
  - Los Angeles, California
  - Montebello, California
  - Sacramento, California
  - Stanford, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Washington D.C, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Camden, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (9):
  - Liverpool, New South Wales
  - St Leonards, New South Wales
  - Wollongong, New South Wales
  - Herston, Queensland
  - Woollongabba, Queensland
  - East Melbourne, Victoria
  - Footscray, Victoria
  - Geelong, Victoria
  - Heidelberg, Victoria
- Austria (2):
  - Linz
  - Vienna
- Belgium (4):
  - Antwerp
  - Brussels
  - Haine-Saint-Paul
  - Leuven
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- France (10):
  - Caen
  - Lille
  - Lyon
  - Montbéliard
  - Nice
  - Pierre-Bénite
  - Rennes
  - Saint-Herblain
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (9):
  - Aachen
  - Berlin
  - Essen
  - Freiberg
  - Hamburg
  - Heidelberg
  - Herne
  - Magdeburg
  - München
- Netherlands (3):
  - Gravenhage
  - Heerlen
  - Rotterdam

REFERENCES:
- [Background] Mehta MP, Shapiro WR, Glantz MJ, Patchell RA, Weitzner MA, Meyers CA, Schultz CJ, Roa WH, Leibenhaut M, Ford J, Curran W, Phan S, Smith JA, Miller RA, Renschler MF. Lead-in phase to randomized trial of motexafin gadolinium and whole-brain radiation for patients with brain metastases: centralized assessment of magnetic resonance imaging, neurocognitive, and neurologic end points. J Clin Oncol. 2002 Aug 15;20(16):3445-53. doi: 10.1200/JCO.2002.07.500. PMID 12177105
- [Background] Carde P, Timmerman R, Mehta MP, Koprowski CD, Ford J, Tishler RB, Miles D, Miller RA, Renschler MF. Multicenter phase Ib/II trial of the radiation enhancer motexafin gadolinium in patients with brain metastases. J Clin Oncol. 2001 Apr 1;19(7):2074-83. doi: 10.1200/JCO.2001.19.7.2074. PMID 11283141
- [Background] Rosenthal DI, Nurenberg P, Becerra CR, Frenkel EP, Carbone DP, Lum BL, Miller R, Engel J, Young S, Miles D, Renschler MF. A phase I single-dose trial of gadolinium texaphyrin (Gd-Tex), a tumor selective radiation sensitizer detectable by magnetic resonance imaging. Clin Cancer Res. 1999 Apr;5(4):739-45. PMID 10213207
- [Background] Magda D, Lepp C, Gerasimchuk N, Lee I, Sessler JL, Lin A, Biaglow JE, Miller RA. Redox cycling by motexafin gadolinium enhances cellular response to ionizing radiation by forming reactive oxygen species. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):1025-36. doi: 10.1016/s0360-3016(01)01810-7. PMID 11704327
- [Background] Miller RA, Woodburn K, Fan Q, Renschler MF, Sessler JL, Koutcher JA. In vivo animal studies with gadolinium (III) texaphyrin as a radiation enhancer. Int J Radiat Oncol Biol Phys. 1999 Nov 1;45(4):981-9. doi: 10.1016/s0360-3016(99)00274-6. PMID 10571206
- See also: National Brain Tumor Foundation — http://www.braintumor.org